CLINICAL TRIAL: NCT05854615
Title: An Observational, Practice-Based, Open Label, Feasibility Study to Observe the Efficacy and Safety of Intramuscular Administration of Stempeucel® in Malaysian Patients With Critical Limb Ischemia (CLI) Due to Buerger's Disease
Brief Title: Efficacy and Safety of Stempeucel® in Patients With Critical Limb Ischemia (CLI) Due to Buerger's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cell Biopeutics Resources Sdn Bhd (Industry)
Collaborators: Stempeutics Research Pvt Ltd (Industry); National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBR-BD-22-003
Record Dates: First submitted 2023-03-30; First posted 2023-05-11 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Critical Limb Ischemia; Buerger's Disease
Keywords: critical limb ischemia; Buerger's disease; bone marrow derived mesenchymal stem cell
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Thromboangiitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stempeucel® (Experimental): Stempeucel® (Ex-vivo cultured MSCs) supplied in 15 ml cryo bags consisting of 200 million or 150 million MSCs, 85% PlasmaLyte-A, 5% HSA and 10% DMSO in a total volume of 15 ml. Following thawing, 35 ml of PlasmaLyte A will be added to the Stempeucel® to make a total volume of 50 ml. The final concentration of components will be 1.5% HSA and 3% DMSO.
  Interventions: Biological: Adult human bone marrow derived, cultured, pooled, allogeneic mesenchymal stromal cells

INTERVENTIONS:
Biological: Adult human bone marrow derived, cultured, pooled, allogeneic mesenchymal stromal cells — • Ex-vivo cultured allogeneic mesenchymal stem cells (MSCs) supplied in cryo-bags consisting of 150 or 200 million, suspended in 50 ml of Plasmalyte A containing 1.5% human serum albumin (HSA) and 3% dimethyl sulfoxide (DMSO).
  Other Names: Stempeucel®

SUMMARY:
The goal of this observational, practice-based feasibility study is to observe the efficacy and safety of intramuscular administration of Stempeucel® in Malaysian patients with critical limb ischemia (CLI) due to Buerger's disease. The main questions it aims to answer are:

* Can intramuscular administration of Stempeucel® reduce symptoms of CLI due to Buerger's disease while improving the healing rate and functional outcomes?
* Does intramuscular administration of Stempeucel® causes any serious adverse events in CLI due to Buerger's disease patients? Study patients will be assessed by the PI before administering the Stempeucel® for any other organ with inflammation. The study patients will also be followed up to the duration of 1 year after study treatment administration for safety and efficacy assessment.

DETAILED DESCRIPTION:
Title: An Observational, Practice-Based, Open Label, Feasibility Study to Observe the Efficacy and Safety of Intramuscular Administration of Stempeucel® in Malaysian Patients with Critical Limb Ischemia (CLI) Due to Buerger's Disease

Study Design: Single arm, practice-based, feasibility study

Study Duration: Estimated duration for the main protocol (e.g. from starts of screening to last subject processed and end of the study) is approximately 18 months

Study Center: Universiti Kebangsaan Malaysia Medical Centre (UKMMMC), Jalan Yaacob Latif, Bandar Tun Razak, 56000 Kuala Lumpur, Wilayah Persekutuan, Malaysia

Objectives: To observe the efficacy and safety of Stempeucel® (adult human bone marrow-derived, cultured, pooled, allogeneic mesenchymal stromal cells) in Malaysian patients with critical limb ischemia (CLI) due to Buerger's disease.

Investigational Medicinal Product

Description

• Ex-vivo cultured allogeneic mesenchymal stem cells (MSCs) supplied in cryo-bags consisting of 150 or 200 million, suspended in 50 ml of Plasmalyte A containing 1.5% human serum albumin (HSA) and 3% dimethyl sulfoxide (DMSO).

Dosage • Dosing of Stempeucel® is based on body weight. The recommended dose is 2 million cells/kg body weight.

Administration

• 40 - 60 injections administered as 0.6 ml/kg (200 million bag) or 0.8 ml/kg (150 million bag) intramuscularly into different points on the muscle. Additional injections of 2 ml (200 million bag) or 3 ml (150 million bag) administered around the ulcer

Number of Subjects 3 patients

Data Analysis

Data Management:

* Electronic case record form (eCRF) will be used for data entry.
* Oracle clinical (or other suitable alternatives with audit trail) will be used for data management.

Statistical Method:

* The SPSS® package (IBM Inc., USA, version 22) will be used for statistical evaluation.
* All patients in the study with relevant efficacy and safety data will be considered for the analysis.
* Efficacy analysis will be done using GEE (Generalized Estimating Equations) method or paired t test as appropriate.
* Adverse events monitored using information voluntarily disclosed by the patients and as observed by the PI will be summarized descriptively by total number of AE(s).
* AEs will be categorized as: all AEs, all treatment-emergent AEs, all severe AEs, treatment-related AEs and severe treatment-related AEs. These events will be reported as appropriate and summarized.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females (willing to use accepted methods of contraception during the course of the study) in the age group of 18-65 years.
2. Buerger's disease as diagnosed by Shionoya criteria
3. Patients should have at least one ulcer (target ulcer): area between 0.5 to 10 cm2 (both inclusive)
4. Ankle Brachial Pressure Index (ABPI) ≤ 0.6. If ABPI is ≥ 1.1 then Toe Brachial Index (TBI) will be performed and TBI should be ≤ 0.5
5. Patients who are able to understand the requirements of the study, and willing to provide voluntary written informed consent, abide by the study requirements, and agree to return for required follow-up visits

Exclusion Criteria:

1. Patients diagnosed with atherosclerotic peripheral arterial disease
2. Patients eligible for surgical or percutaneous revascularization
3. Patients with a history of participating in another stem cell trial or therapy within 3 months
4. Patients who are unsuitable to participate the clinical trial as determined by investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in ischemic rest pain | Screening (Day -14 to -1), Day 30, 90, 180 and 360
  Change in visual analog score (VAS) compared to screening
Change in size of the ulcer | Screening (Day -14 to -1), Day 30, 90, 180 and 360
  Change in size of the ulcer compared to screening
Change in ankle brachial pressure index (ABPI) | Screening (Day -14 to -1), Day 30, 90, 180 and 360
  Change in ankle brachial pressure index (ABPI) compared to screening
Change in total walking distance | Screening (Day -14 to -1), Day 30, 90, 180 and 360
  Change in total walking distance on a treadmill compared to screening
Change in major amputation-free survival | Screening (Day -14 to -1), Day 30, 90, 180 and 360
  Change in amputation-free survival compared to screening
Change in angiogenesis | Screening (Day -14 to -1), Day 180
  Change in angiogenesis measured by digital subtraction angiogram (DSA) compared to screening

SECONDARY OUTCOMES:
The type of AE(s), number of AE(s) and proportion of patients with AE(s) | Screening (Day -14 to -1)
  AE(s) will be monitored and recorded as voluntarily disclosed by the patients and as observed by the investigator throughout the study
Incidence of abnormal laboratory test results (serum chemistry, haematology, liver function test) | Screening (Day -14 to -1), Day 7, 30, 90, 180 and 360
  The following lab tests will be conducted: serum chemistry, haematology, liver function test. In case of abnormal results, they shall be recorded as an adverse event or excluded from study (screening).
Incidence of abnormal urine test results | Screening (Day -14 to -1), Day 180
  Urine test will be conducted. In case of abnormal results, they shall be recorded as an adverse event or excluded from study (screening).
Incidence of abnormal TNF-α | Screening (Day -14 to -1), Day 7 and 30
  TNF-α test will be conducted. In case of abnormal results, they shall be recorded as an adverse event or excluded from study (screening).
Incidence of abnormal vital signs | Screening (Day -14 to -1), Baseline, Day 7, 30, 90, 180 and 360
  The following assessments will be conducted: blood pressure, heart rate, respiratory rate and temperature. In case of abnormal results, they shall be recorded as an adverse event or excluded from study (screening).
Incidence of abnormal physical examination | Screening (Day -14 to -1), Baseline, Day 7, 30, 90, 180 and 360
  The following examinations will be conducted: visual, heart, lungs, abdomen, nervous system, muscoskeletal system and etc. In case of abnormal conditions, they shall be recorded as an adverse event or excluded from study (screening).
Incidence of abnormal ECG parameters | Screening (Day -14 to -1), Baseline, Day 7, 30, 90, 180 and 360
  The following assessments will be conducted: 12 lead ECG recordings with long Lead II, and two-dimensional echocardiography (2D ECHO; if needed). In case of abnormal conditions, they shall be recorded as an adverse event or excluded from study (screening).
Incidence of abnormal chest condition | Screening (Day -14 to -1), Day 180
  Chest x-ray will be conducted. In case of abnormal conditions, they shall be recorded as an adverse event or excluded from study (screening).

CONTACTS AND LOCATIONS:
Overall Officials: Hanafiah Harunarashid, MS, Principal Investigator — National University of Malaysia
Locations (1):
- Hospital Canselor Tunku Mukhriz, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haugen S, Casserly IP, Regensteiner JG, Hiatt WR. Risk assessment in the patient with established peripheral arterial disease. Vasc Med. 2007 Nov;12(4):343-50. doi: 10.1177/1358863X07083278. PMID 18048472
- [Background] Sprengers RW, Lips DJ, Moll FL, Verhaar MC. Progenitor cell therapy in patients with critical limb ischemia without surgical options. Ann Surg. 2008 Mar;247(3):411-20. doi: 10.1097/SLA.0b013e318153fdcb. PMID 18376183
- [Background] Dormandy J, Heeck L, Vig S. The fate of patients with critical leg ischemia. Semin Vasc Surg. 1999 Jun;12(2):142-7. PMID 10777241
- [Background] Gottsater A. Managing risk factors for atherosclerosis in critical limb ischaemia. Eur J Vasc Endovasc Surg. 2006 Nov;32(5):478-83. doi: 10.1016/j.ejvs.2006.03.007. Epub 2006 Apr 24. PMID 16631394
- [Background] Schiavetta A, Maione C, Botti C, Marino G, Lillo S, Garrone A, Lanza L, Pagliari S, Silvestroni A, Signoriello G, Sica V, Cobellis G. A phase II trial of autologous transplantation of bone marrow stem cells for critical limb ischemia: results of the Naples and Pietra Ligure Evaluation of Stem Cells study. Stem Cells Transl Med. 2012 Jul;1(7):572-8. doi: 10.5966/sctm.2012-0021. Epub 2012 Jul 6. PMID 23197862
- [Background] Fadini GP, Agostini C, Avogaro A. Autologous stem cell therapy for peripheral arterial disease meta-analysis and systematic review of the literature. Atherosclerosis. 2010 Mar;209(1):10-7. doi: 10.1016/j.atherosclerosis.2009.08.033. Epub 2009 Aug 21. PMID 19740466
- [Background] Conte MS, Geraghty PJ, Bradbury AW, Hevelone ND, Lipsitz SR, Moneta GL, Nehler MR, Powell RJ, Sidawy AN. Suggested objective performance goals and clinical trial design for evaluating catheter-based treatment of critical limb ischemia. J Vasc Surg. 2009 Dec;50(6):1462-73.e1-3. doi: 10.1016/j.jvs.2009.09.044. Epub 2009 Nov 7. PMID 19897335
- [Background] Marston WA, Davies SW, Armstrong B, Farber MA, Mendes RC, Fulton JJ, Keagy BA. Natural history of limbs with arterial insufficiency and chronic ulceration treated without revascularization. J Vasc Surg. 2006 Jul;44(1):108-114. doi: 10.1016/j.jvs.2006.03.026. PMID 16828434
- [Background] Gupta NK, Armstrong EJ, Parikh SA. The current state of stem cell therapy for peripheral artery disease. Curr Cardiol Rep. 2014 Feb;16(2):447. doi: 10.1007/s11886-013-0447-2. PMID 24414120
- [Background] Tachi Y, Fukui D, Wada Y, Koshikawa M, Shimodaira S, Ikeda U, Amano J. Changes in angiogenesis-related factors in serum following autologous bone marrow cell implantation for severe limb ischemia. Expert Opin Biol Ther. 2008 Jun;8(6):705-12. doi: 10.1517/14712598.8.6.705. PMID 18476781
- [Background] Amann B, Luedemann C, Ratei R, Schmidt-Lucke JA. Autologous bone marrow cell transplantation increases leg perfusion and reduces amputations in patients with advanced critical limb ischemia due to peripheral artery disease. Cell Transplant. 2009;18(3):371-80. doi: 10.3727/096368909788534942. Epub 2009 Apr 2. PMID 19500466
- [Background] Molavi B, Zafarghandi MR, Aminizadeh E, Hosseini SE, Mirzayi H, Arab L, Baharvand H, Aghdami N. Safety and Efficacy of Repeated Bone Marrow Mononuclear Cell Therapy in Patients with Critical Limb Ischemia in a Pilot Randomized Controlled Trial. Arch Iran Med. 2016 Jun;19(6):388-96. PMID 27293053
- [Background] Liang TW, Jester A, Motaganahalli RL, Wilson MG, G'Sell P, Akingba GA, Fajardo A, Murphy MP. Autologous bone marrow mononuclear cell therapy for critical limb ischemia is effective and durable. J Vasc Surg. 2016 Jun;63(6):1541-5. doi: 10.1016/j.jvs.2016.01.022. Epub 2016 Mar 23. PMID 27021379
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Lawall H, Bramlage P, Amann B. Stem cell and progenitor cell therapy in peripheral artery disease. A critical appraisal. Thromb Haemost. 2010 Apr;103(4):696-709. doi: 10.1160/TH09-10-0688. Epub 2010 Feb 19. PMID 20174766
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076
- [Background] Shi Q, Rafii S, Wu MH, Wijelath ES, Yu C, Ishida A, Fujita Y, Kothari S, Mohle R, Sauvage LR, Moore MA, Storb RF, Hammond WP. Evidence for circulating bone marrow-derived endothelial cells. Blood. 1998 Jul 15;92(2):362-7. PMID 9657732
- [Background] Tateishi-Yuyama E, Matsubara H, Murohara T, Ikeda U, Shintani S, Masaki H, Amano K, Kishimoto Y, Yoshimoto K, Akashi H, Shimada K, Iwasaka T, Imaizumi T; Therapeutic Angiogenesis using Cell Transplantation (TACT) Study Investigators. Therapeutic angiogenesis for patients with limb ischaemia by autologous transplantation of bone-marrow cells: a pilot study and a randomised controlled trial. Lancet. 2002 Aug 10;360(9331):427-35. doi: 10.1016/S0140-6736(02)09670-8. PMID 12241713
- [Background] Lu Y, Wang Z, Zhu M. Human bone marrow mesenchymal stem cells transfected with human insulin genes can secrete insulin stably. Ann Clin Lab Sci. 2006 Spring;36(2):127-36. PMID 16682507
- [Background] Oswald J, Boxberger S, Jorgensen B, Feldmann S, Ehninger G, Bornhauser M, Werner C. Mesenchymal stem cells can be differentiated into endothelial cells in vitro. Stem Cells. 2004;22(3):377-84. doi: 10.1634/stemcells.22-3-377. PMID 15153614
- [Background] Tse WT, Pendleton JD, Beyer WM, Egalka MC, Guinan EC. Suppression of allogeneic T-cell proliferation by human marrow stromal cells: implications in transplantation. Transplantation. 2003 Feb 15;75(3):389-97. doi: 10.1097/01.TP.0000045055.63901.A9. PMID 12589164
- [Background] Di Nicola M, Carlo-Stella C, Magni M, Milanesi M, Longoni PD, Matteucci P, Grisanti S, Gianni AM. Human bone marrow stromal cells suppress T-lymphocyte proliferation induced by cellular or nonspecific mitogenic stimuli. Blood. 2002 May 15;99(10):3838-43. doi: 10.1182/blood.v99.10.3838. PMID 11986244
- [Background] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814
- [Background] Muraglia A, Cancedda R, Quarto R. Clonal mesenchymal progenitors from human bone marrow differentiate in vitro according to a hierarchical model. J Cell Sci. 2000 Apr;113 ( Pt 7):1161-6. doi: 10.1242/jcs.113.7.1161. PMID 10704367
- [Background] Reyes M, Verfaillie CM. Characterization of multipotent adult progenitor cells, a subpopulation of mesenchymal stem cells. Ann N Y Acad Sci. 2001 Jun;938:231-3; discussion 233-5. doi: 10.1111/j.1749-6632.2001.tb03593.x. PMID 11458512
- [Background] Devine SM, Bartholomew AM, Mahmud N, Nelson M, Patil S, Hardy W, Sturgeon C, Hewett T, Chung T, Stock W, Sher D, Weissman S, Ferrer K, Mosca J, Deans R, Moseley A, Hoffman R. Mesenchymal stem cells are capable of homing to the bone marrow of non-human primates following systemic infusion. Exp Hematol. 2001 Feb;29(2):244-55. doi: 10.1016/s0301-472x(00)00635-4. PMID 11166464
- [Background] Bhatia R, Hare JM. Mesenchymal stem cells: future source for reparative medicine. Congest Heart Fail. 2005 Mar-Apr;11(2):87-91; quiz 92-3. doi: 10.1111/j.1527-5299.2005.03618.x. PMID 15860974
- [Background] Shintani S, Murohara T, Ikeda H, Ueno T, Sasaki K, Duan J, Imaizumi T. Augmentation of postnatal neovascularization with autologous bone marrow transplantation. Circulation. 2001 Feb 13;103(6):897-903. doi: 10.1161/01.cir.103.6.897. PMID 11171801
- [Background] Kamihata H, Matsubara H, Nishiue T, Fujiyama S, Tsutsumi Y, Ozono R, Masaki H, Mori Y, Iba O, Tateishi E, Kosaki A, Shintani S, Murohara T, Imaizumi T, Iwasaka T. Implantation of bone marrow mononuclear cells into ischemic myocardium enhances collateral perfusion and regional function via side supply of angioblasts, angiogenic ligands, and cytokines. Circulation. 2001 Aug 28;104(9):1046-52. doi: 10.1161/hc3501.093817. PMID 11524400
- [Background] Iba O, Matsubara H, Nozawa Y, Fujiyama S, Amano K, Mori Y, Kojima H, Iwasaka T. Angiogenesis by implantation of peripheral blood mononuclear cells and platelets into ischemic limbs. Circulation. 2002 Oct 8;106(15):2019-25. doi: 10.1161/01.cir.0000031332.45480.79. PMID 12370229 (Retraction: PMID 23704253 Circulation. 2013 Jun 11;127(23):e842)
- [Background] Kalka C, Masuda H, Takahashi T, Kalka-Moll WM, Silver M, Kearney M, Li T, Isner JM, Asahara T. Transplantation of ex vivo expanded endothelial progenitor cells for therapeutic neovascularization. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3422-7. doi: 10.1073/pnas.97.7.3422. PMID 10725398
- [Background] Wu Y, Chen L, Scott PG, Tredget EE. Mesenchymal stem cells enhance wound healing through differentiation and angiogenesis. Stem Cells. 2007 Oct;25(10):2648-59. doi: 10.1634/stemcells.2007-0226. Epub 2007 Jul 5. PMID 17615264
- [Background] Mahmud N, Pang W, Cobbs C, Alur P, Borneman J, Dodds R, Archambault M, Devine S, Turian J, Bartholomew A, Vanguri P, Mackay A, Young R, Hoffman R. Studies of the route of administration and role of conditioning with radiation on unrelated allogeneic mismatched mesenchymal stem cell engraftment in a nonhuman primate model. Exp Hematol. 2004 May;32(5):494-501. doi: 10.1016/j.exphem.2004.02.010. PMID 15145218
- [Background] Bhattacharya V, McSweeney PA, Shi Q, Bruno B, Ishida A, Nash R, Storb RF, Sauvage LR, Hammond WP, Wu MH. Enhanced endothelialization and microvessel formation in polyester grafts seeded with CD34(+) bone marrow cells. Blood. 2000 Jan 15;95(2):581-5. PMID 10627466
- [Background] Ikenaga S, Hamano K, Nishida M, Kobayashi T, Li TS, Kobayashi S, Matsuzaki M, Zempo N, Esato K. Autologous bone marrow implantation induced angiogenesis and improved deteriorated exercise capacity in a rat ischemic hindlimb model. J Surg Res. 2001 Apr;96(2):277-83. doi: 10.1006/jsre.2000.6080. PMID 11266284
- [Background] Hirata K, Li TS, Nishida M, Ito H, Matsuzaki M, Kasaoka S, Hamano K. Autologous bone marrow cell implantation as therapeutic angiogenesis for ischemic hindlimb in diabetic rat model. Am J Physiol Heart Circ Physiol. 2003 Jan;284(1):H66-70. doi: 10.1152/ajpheart.00547.2002. Epub 2002 Sep 19. PMID 12388231
- [Background] Gupta PK, Chullikana A, Parakh R, Desai S, Das A, Gottipamula S, Krishnamurthy S, Anthony N, Pherwani A, Majumdar AS. A double blind randomized placebo controlled phase I/II study assessing the safety and efficacy of allogeneic bone marrow derived mesenchymal stem cell in critical limb ischemia. J Transl Med. 2013 Jun 10;11:143. doi: 10.1186/1479-5876-11-143. PMID 23758736
- [Background] Gupta PK, Krishna M, Chullikana A, Desai S, Murugesan R, Dutta S, Sarkar U, Raju R, Dhar A, Parakh R, Jeyaseelan L, Viswanathan P, Vellotare PK, Seetharam RN, Thej C, Rengasamy M, Balasubramanian S, Majumdar AS. Administration of Adult Human Bone Marrow-Derived, Cultured, Pooled, Allogeneic Mesenchymal Stromal Cells in Critical Limb Ischemia Due to Buerger's Disease: Phase II Study Report Suggests Clinical Efficacy. Stem Cells Transl Med. 2017 Mar;6(3):689-699. doi: 10.5966/sctm.2016-0237. Epub 2016 Oct 5. PMID 28297569
- [Background] Bura A, Planat-Benard V, Bourin P, Silvestre JS, Gross F, Grolleau JL, Saint-Lebese B, Peyrafitte JA, Fleury S, Gadelorge M, Taurand M, Dupuis-Coronas S, Leobon B, Casteilla L. Phase I trial: the use of autologous cultured adipose-derived stroma/stem cells to treat patients with non-revascularizable critical limb ischemia. Cytotherapy. 2014 Feb;16(2):245-57. doi: 10.1016/j.jcyt.2013.11.011. PMID 24438903
- [Background] Wester T, Jorgensen JJ, Stranden E, Sandbaek G, Tjonnfjord G, Bay D, Kolleros D, Kroese AJ, Brinchmann JE. Treatment with autologous bone marrow mononuclear cells in patients with critical lower limb ischaemia. A pilot study. Scand J Surg. 2008;97(1):56-62. doi: 10.1177/145749690809700108. PMID 18450207
- [Background] Debin L, Youzhao J, Ziwen L, et al. Autologous transplantation of bone marrow mesenchymal stem cells on diabetic patients with lower limb ischemia. Journal of Medical Colleges of PLA. 2008; 23(2): 106-155. doi: 10.1016/S1000-1948(08)60031-3
- [Background] Idei N, Soga J, Hata T, Fujii Y, Fujimura N, Mikami S, Maruhashi T, Nishioka K, Hidaka T, Kihara Y, Chowdhury M, Noma K, Taguchi A, Chayama K, Sueda T, Higashi Y. Autologous bone-marrow mononuclear cell implantation reduces long-term major amputation risk in patients with critical limb ischemia: a comparison of atherosclerotic peripheral arterial disease and Buerger disease. Circ Cardiovasc Interv. 2011 Feb 1;4(1):15-25. doi: 10.1161/CIRCINTERVENTIONS.110.955724. Epub 2011 Jan 4. PMID 21205941
- [Background] Rasmusson I. Immune modulation by mesenchymal stem cells. Exp Cell Res. 2006 Jul 15;312(12):2169-79. doi: 10.1016/j.yexcr.2006.03.019. Epub 2006 Apr 24. PMID 16631737
- [Background] ICH Topic E 2 A:Clinical Safety Data Management: Definitions and Standards for Expedited Reporting-(CPMP/ICH/377/95)
- [Background] Central Drugs Standard Control Organization, Directorate General of Health Services, Ministry of Health & Family Welfare, Govt. of India. Draft Guidelines on Audio-Visual Recording of Informed Consent Process in Clinical Trial. 2014. [cited 2016 Jul 29]. Available from: http://www.cdsco.nic.in/writereaddata/Guidance_for_AV%20Recording_09.January.14.pdf.
- [Background] ClinicalTrials.gov. Identifier NCT01257776, Human Adipose Derived Mesenchymal Stem Cells for Critical Limb Ischemia (CLI) in Diabetic Patients. Available from: http://clinicaltrials.gov/ct2/show/NCT01079403

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT05854615/Prot_SAP_000.pdf